CLINICAL TRIAL: NCT01216566
Title: Computerized Mobilization of the Cervical Spine Utilizing the Occiflex Device for the Treatment of Chronic Neck Pain
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Headway Ltd. (Unknown)
Responsible Party: Yaron River, MD, Dept. of Neurology, Hillel Yaffe Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYMC-0030-10
Record Dates: First submitted 2010-06-01; First posted 2010-10-07 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I. Patients with chronic neck pain (Experimental)
  Interventions: Device: Occiflex Device

INTERVENTIONS:
Device: Occiflex Device — This device is a computerized robotic platform that allows continuous mobilization of the cervical spine in a three dimensional space. The patients undergoes biweekly 20 minute therapeutic session for 6 weeks

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of the Occiflex device in the treatment of neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic neck pain: post-whiplash injury, myofacial pain, cervical facet joint disease and idiopathic chronic neck pain

Exclusion Criteria:

* Radiculopathy
* Myelopathy
* Cerebral vascular disease
* Malignancy
* Osteoporosis
* Cervical disc herniation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-04 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Safety of computerized continuous mobilization of the cervical spine | one year

SECONDARY OUTCOMES:
Efficacy of computerized mobilization of treatment of patients with chronic neck pain | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel